CLINICAL TRIAL: NCT00974454
Title: Research on Effect of TCM on Immune Reconstitution of HIV/AIDS Patients After HAART
Brief Title: Research on Effect of Traditional Chinese Medicine (TCM) on Immune Reconstitution of HIV/AIDS Patients After Highly Active Antiretroviral Therapy (HAART)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: WANG, Jie/Professor, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09.07.16-1
Record Dates: First submitted 2009-09-09; First posted 2009-09-10 (Estimated); Last update posted 2009-10-29 (Estimated); Status verified 2009-09

CONDITIONS: Acquired Immune Deficiency Syndrome Virus; HIV Infections
Keywords: AIDS; complementary therapies; treatment experienced
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fuzheng 2 (Active Comparator): Immunity 2 (Fuzheng 2), 6.25g twice a day, half an hour before breakfast and dinner, mixing with water, for six successive cycles of 30 days.
  Interventions: Drug: Fuzheng 2
- Placebo (Placebo Comparator): Placebo, 6.25g twice a day, half an hour before breakfast and dinner, mixing with water, for six successive cycles of 30 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fuzheng 2 — Immunity 2 (Fuzheng 2), 6.25g twice a day, half an hour before breakfast and dinner, mixing with water, for six successive cycles of 30 days.
  Arms: Fuzheng 2
Drug: Placebo — Placebo, 6.25g twice a day, half an hour before breakfast and dinner, mixing with water, for six successive cycles of 30 days.
  Arms: Placebo

SUMMARY:
Chinese prescriptions can inhibit viral replication according to the course of viral replication, and the effects is similar to the effect of HAART, and even better than the anti-viral and immune reconstitution of HAART due to its effect on improve immune system function. Over the past decades, many researchers have screened the effective Chinese medicines to treat AIDS.

DETAILED DESCRIPTION:
* There is no record of AIDS in Chinese medicine, modern clinicians hold that AIDS is linked to TCM theory according to its pathogenesis, character of onset and clinical manifestations. As early as more than 2000 years ago, there were records of immune function in TCM. 2 TCM books recorded that "keep vital Qi, the evil will not invade the body "and" the invasion of evil is caused by the deficiency of vital Qi. Vital Qi summarizes the normal immune system function. Vital Qi is the basic material and physiological function which can eliminate the evil, regulating yin and yang and protect the body.
* And this is in accordance with defense, homeostasis and surveillance of immune system in western medicine. The knowledge of immunology has guided medical practice in China for more than two thousand years. In response to a variety of immune diseases, there are various immunotherapy such as Yiqi Fuzheng immunotherapy, reinforce kidney therapy, huoxuehuayu therapy and heat-clearing and detoxifying therapy. Throughout the course of AIDS, the evil (HIV) exists and the vital Qi is turning weak gradually. If we adopted a number of intervention measures to assist the body's Vital Qi, Vital Qi will be strengthened and the evil will be weakened. Therefore, TCM will play an important role in improving immune function.
* Chinese prescriptions can inhibit viral replication according to the course of viral replication, and the effects is similar to the effect of HAART, and even better than the anti-viral and immune reconstitution of HAART due to its effect on improve immune system function. Over the past decades, many researchers have screened the effective Chinese medicines to treat AIDS.

Researchers screened single Chinese herbs, some extract and the effective components of Chinese medicine and prescriptions. Some study the role of its anti-HIV, some study the role of its regulating immunization function. The former studies have shown that immunization 2 (Fuzheng 2) has wide effect on immune system and it can activate the reticuloendothelial system, macrophage phagocytes and lymphocyte transformation. And it can relieve disorders, imbalance of the immune system caused by HIV infection.

* In addition, this prescription can inhibit HIV reverse transcription polymerase enzyme and virus-induced syncytium formation, protect virus-infected cells, and inhibit virus replication in HIV-1 infected cells.
* Through the clinical trials, we will evaluate the effect of immune 2 (Fuzheng 2) on immune reconstitution of adult HIV/AIDS patients who have received HAART.

ELIGIBILITY:
Inclusion Criteria:

* HIV antibody-positive, confirmed by Western Blot test
* HIV antibody-positive, confirmed by Western Blot test
* HAART ≥ 12 months
* CD 4 count increased by <100 cells / ul
* HIV RNA <50 c / ml (bDNA);
* Age ≥ 18 years old and ≤ 70 years old
* Voluntary participated in this study, signed informed consent form, and could be followed-up

Exclusion Criteria:

* Serious opportunistic infections were not brought under control (Pneumocystis carinii pneumonia, meningitis, esophageal candidiasis, lymphoma, toxoplasma encephalopathy, tuberculosis, etc.) before the experiment
* Participated in clinical trials of other drugs within one month before the experiment
* Received immunomodulatory treatment within one month before the experiment
* WBC <2 × 10 9 / L, N <1.0 × 10 9 / L, Hb <90g / L, PLT <75 × 10 9 / L,liver and kidney dysfunction (AST, ALT, T-BIL ≥2 times of upper limit of the reference value or creatinine ≥ 2 times of the upper limit of reference value)
* Patients with pancreatitis or active gastric ulcer
* Patients with obvious active diseases in respiratory system, digestive system, circulatory system, blood system, neuroendocrine system, or genitourinary system diseases
* Persons suffering from autoimmune diseases
* Cancer patients which need chemotherapy
* Pregnant or lactating women, and did not use safe contraceptive measures for women of child-bearing age, as well as the male that can not take a reasonable method of contraception in trial period
* Hypersensitive people
* Patients with dysgnosia or language barriers, which can not fully understand the test or cooperate well

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-04 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Peripheral blood CD3+ CD4+ counts | 6 months

SECONDARY OUTCOMES:
Immune reconstitution efficiency | 6 months
Viral load | 6 months
Clinical symptoms and signs | 6 months
KPS score | 6 months
Quality of life score | 6 months
Side effects of HAART | 6 months
Safety evaluation | 6 months
Economic evaluation | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jie WANG, MD, Study Chair — Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- Guang'anmen Hospital of China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China